CLINICAL TRIAL: NCT01117558
Title: The Risk of Metabolic Syndrome and Cardiovascular Disease in Women With Polycystic Ovary Syndrome.
Brief Title: Study of Metabolism and Cardiovascular Disease(CVD) in Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-98010
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS,; DM,; Hypertension,; CVD
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
PCOS is the most common endocrine disorder in reproductive women. It is estimated that 5 to 10% of women of reproductive age have PCOS. One of the major diagnostic criteria of PCOS was chronic anovulation which lead to irregular menstruation, amenorrhea, and infertility; the other diagnostic criteria was hyperandrogenism which lead to hirsutism, acne and alopecia. Furthermore, PCOS is thought as a metabolic disorder, the long-term consequence of PCOS were diabetes mellitus and cardiovascular disease, which are potentially dangerous in women health. Early diagnosis and prevention is very important to the PCOS patients.

Obesity is the most potential risk of threat to health of populations. There is a major impact of obesity on the PCOS related disorders. Insulin resistance and distribution of adipose tissue were thought to be the important risk factors of cardiovascular and metabolic syndrome.

To treat PCOS patients properly,Wan-Fang hospital had established a specific medical team. The investigators recently published in "Fertility and Sterility" about the clinical presentation of androgen excess in Taiwanese women. Hirsutism is much less prevalence in Taiwanese PCOS women than that previous reported in the Western women. It is important to know that some clinical presentation of PCOS might have ethic variance. Insulin resistance was reported as another candidate that might have ethic variance.The investigators had reported about 40% women in PCOS women were obese, it is similar with previous literature reported. Obesity is a major factor that could be controlled during the treatment of PCOS.Weight reduction is one of our methods in PCOS treatment. The progressive results for obese PCOS women would be facing the risks of diabetes and metabolic syndrome.The investigators thought like to evaluate the benefit of weight reduction program to the prognosis of obese women with PCOS. Furthermore, it is known that Endothelial progenitor cells (EPC) be an early marker of cardiovascular disease, the investigators would like to know the role of EPC to predict metabolic syndrome in women with PCOS. Wan-Fang hospital has a professional team in PCOS treatment and research which including gynecological endocrinologist, cardiologist, medical endocrinologist, specialist in weight reduction. This team had been working well for more that 4 years.

The investigators hope that they can make a contribution to the study and treatment of PCOS in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* PCOM by ultrasound Diagnosis
* Anovulation, Oligo menses
* Hyperandrogenism

Exclusion Criteria:

* Women who had been diagnosed with other etiology that should be excluded in PCOS diagnosis, such as hyperprolactinemia, hypogonadotropic hypogonadism, premature ovarian failure, congenital adrenal hyperplastic, androgen-secreting tumor, Cushing's syndrome, disorders of uterus (such as Asherman's syndrome, Mullerian agenesis), chromosomal anomalies (such as Turner syndrome).
* Women who did not have sufficient clinical or biochemical records.
* Girls who had menarche at <3 years of age and women who were >40 years of age.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic Ovary Syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
obesity | prospectively recruited from June 1, 2009 to September 31, 2010.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taipei, Taiwan